CLINICAL TRIAL: NCT02415582
Title: Effects of Different Exercises on Post-Exercise Blood Pressure in Elderly Hypertensive: A Cross-Over Randomized Clinical Trial
Brief Title: Post-Exercise Hypotension in Elderly Hypertensive Men
Acronym: HPE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital de Clinicas de Porto Alegre (Other)
Collaborators: Federal University of Rio Grande do Sul (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: 130484
Record Dates: First submitted 2015-04-09; First posted 2015-04-14 (Estimated); Last update posted 2018-05-31 (Actual); Status verified 2015-08

CONDITIONS: Hypertension
Keywords: Hypertension; Bloodpressure; Post-exercise hypotension; Combined exercise; Aerobic exercise; Resistance exercise; Aging; Elderly; Ambulatory blood pressure monitoring
MeSH Terms: conditions — Hypertension; Post-Exercise Hypotension | interventions — Exercise

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Aerobic exercise (Experimental): Aerobic exercise on treadmill at 65-70% of the heart rate reserve during a session.
  Interventions: Other: Aerobic exercise
- Combined exercises (Experimental): A session combines resistance and aerobic exercises, with aerobic exercise on treadmill at 65-70% of the heart rate reserve, followed by 60 minutes for cardiorespiratory recovery, and resistance exercise.
  Interventions: Other: Combined exercises
- Control (Sham Comparator): Participants do not exercise and remain sitting for 45 minutes
  Interventions: Other: Control

INTERVENTIONS:
Other: Aerobic exercise — Aerobic exercise on treadmill
  Arms: Aerobic exercise
Other: Combined exercises — Combined resistance and aerobic exercise
  Arms: Combined exercises
Other: Control — 45 minutes resting sitting
  Arms: Control

SUMMARY:
The purpose of this study is to compare the effects of two exercise protocols on post-exercise blood pressure versus a control group in elderly hypertensive men. Participants are allocated to all groups: control group and two experimental exercise protocols, in a random order. In the control group, participants remain resting sitting, and, in the exercise protocols, participants practice exercise bouts of aerobic exercise or a combination of resistance and aerobic exercises. In order to standardize baseline conditions, before the sessions subjects remain sitting quietly for 20 minutes. After each exercise protocol, participants have 60 minutes for recovery and, simultaneously, they have BP measured every 5 minutes. After the exercise sessions or control, an equipment for 24 hours ambulatory BP monitoring is installed in every participant.

DETAILED DESCRIPTION:
Hypertension has high prevalence and low rate of control, and is a major modifiable risk factor and public health problem. Regular physical exercise is a relevant non-pharmacological option for prevention and treatment of hypertension. Several studies demonstrated a reduction in blood pressure (BP) following different exercise protocols, and the decrease may be the result of the summation of hypotensive effects that occur in the hours following the workout. The reduction resulting from a single exercise session is called post-exercise hypotension (PEH) and has been investigated among hypertensive subjects. However, to achieve clinical relevance the PEH should reach a significant magnitude and the reduction should be sustained for a longer period.

Previous studies showed the positive effects of aerobic exercise on post-exercise hypotension in hypertensive subjects. However, there is lacking evidence regarding the effects of a single session of aerobic and resistance exercise combined, and the duration of its effect in 24 hours blood pressure in elderly hypertensive subjects.

The study is an open, crossover randomized clinical trial, with elderly men allocated to three arms, in a random order:

* Aerobic training session
* Combined resistance training and aerobic session
* Control session

After each exercise session, participants have 60 minutes for recovery, performed in the sitting position, with BP measurements every 5 minutes. In addition, participants have measured BP using 24h ambulatory BP monitoring. At the end of the trial, participants will have completed all three experimental protocols: a non-exercise control session, of sitting rest, and two exercise bouts, one of aerobic exercise and a combined resistance and aerobic exercise, with seven days of washout period among sessions. All experiments will be conducted at the same time of day to account for diurnal BP variation. Before the experimental sessions, participants are enrolled in three pre-intervention tests: a familiarization session, cardiopulmonary exercise testing and one maximum repetition strength test (1RM). The aerobic sessions last for 45 minutes, as well as the resistance exercises, and the session of control.

ELIGIBILITY:
Inclusion Criteria:

* Essential hypertension grade 1 - 2 with or without medical treatment:

resting systolic blood pressure (SBP) ≥ 140 mmHg or diastolic blood pressure (DBP) ≥ 90 mmHg

Exclusion Criteria:

* Smoking;
* Bone, joint, or muscle problems that could limit the performance of the exercises.
* BMI ≥ 30 kg/m2
* Heart Attack in the last year

Ages: 60 Years to 70 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2014-03; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Ambulatory Blood Pressure Monitoring | 24 hours
  Ambulatory blood pressure monitoring following experimental protocols

SECONDARY OUTCOMES:
Office Blood Pressure | 1 hour
  Post exercise blood pressure during 60 minutes after experimental sessions

CONTACTS AND LOCATIONS:
Overall Officials: Sandra C Fuchs, PhD, Principal Investigator — Hospital de Clinicas de Porto Alegre
Locations (1):
- Hospital de Clinicas de Porto Alegre, Porto Alegre, Rio Grande do Sul, Brazil